CLINICAL TRIAL: NCT03085290
Title: Allogeneic Versus Autologous Serum Eye Drops: a Double-blind Randomized Cross Over Trial
Brief Title: Allogeneic Versus Autologous Serum Eye Drops
Acronym: AVAnS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sanquin Research & Blood Bank Divisions (Other)
Collaborators: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NL53068.091.15
Record Dates: First submitted 2017-03-02; First posted 2017-03-21 (Actual); Last update posted 2019-04-04 (Actual); Status verified 2019-04

CONDITIONS: Dry Eye Syndrome
Keywords: dry eye syndrome; serum eye drops
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): Subjects assigned to this arm will receive autologous serum eye drops first, followed by a washout period and then allogeneic serum eye drops.
  Interventions: Other: Autologous serum eye drops; Other: Allogeneic serum eye drops
- Group B (Experimental): Subjects assigned to this arm will receive allogeneic serum eye drops first, followed by a washout period and then autologous serum eye drops.
  Interventions: Other: Autologous serum eye drops; Other: Allogeneic serum eye drops

INTERVENTIONS:
Other: Autologous serum eye drops — Autologous serum eye drop doses will be 6 times daily in each eye
Other: Allogeneic serum eye drops — Allogeneic serum eye drop doses will be 6 times daily in each eye

SUMMARY:
Serum eye drops (SEDs) are used to treat patients with extreme dry eyes and other corneal defects. Serum is used in severe ophthalmic cases where conventional eye drops (artificial tears) have insufficient effect. The use of SEDs in dry eye patients usually has a rapid effect. Most patients claim the effect to be instantaneous, and all symptoms improve within 48 hours.

There is evidence suggesting that substances in serum may help in the healing of epithelial defects, such as epidermal growth factor, fibroblast growth factor, fibronectin, and/or vitamin A. However, the precise serum factor responsible for alleviating the patient's complaints is currently not known. Commonly, autologous SEDs are used, but they are replaced more and more by allogeneic SEDs prepared from donor serum.

Allogeneic SED are derived from healthy voluntary, non-remunerated male donors with blood group AB. The use of allogeneic SED could provide blood bank controlled quality, a safer product in larger quantities that is quickly available for each patient.

No double-blind randomized trials are known to exist to detect a difference in result between the effect of allogeneic SED or autologous SED. This pilot study is intended to obtain insight in the ability of autologous and allogeneic SEDs to improve patient dry eye sensation. Our hypothesis is that autologous SEDs (in a 1:1 dilution with saline) result in an improvement of the patient dry eye sensation, while allogeneic SEDs (in a 1:1 dilution with saline) do not.

DETAILED DESCRIPTION:
Serum eye drops (SEDs) are used to treat patients with dry eyes and other diseases, like corneal defects. SEDs are used in ophthalmic cases where conventional eye drops have insufficient effect. The use of SEDs in dry eye patients usually has a rapid effect. Most patients claim the effect to be instantaneous and all symptoms improve by 48 hours [1].

There is evidence suggesting that serum may enhance corneal epithelial healing [2]. Some biologically active substances are thought to contribute to the positive effects, like epidermal growth factor, fibroblast growth factor, fibronectin, and vitamin A.

Autologous SEDs are used internationally on a regular basis, and allogeneic SEDs are becoming increasingly popular. In the Netherlands, only autologous SEDs are in use.

Obtaining autologous SED is an organizational burden. Patient-related problems are old age, travelling, or travelling with low vision and sometimes immobility due to other diseases. Sometimes venipuncture is impossible due to poor access. Medical conditions such as inability to donate large amounts of whole blood due to previous cerebrovascular accidents or cardiovascular disease, anemia, or use of certain medication may prevent collection of blood for SEDs. Patients affected with hematological diseases, bacterial, viral or fungal infections are also unsuitable for production of autologous SEDs. In 2.3% of donors for preparing autologous SEDs, a systemic infection can be detected [3]. In the UK, use of autologous SED is restricted largely due to cost [4]. Logistically, it is a problem that it takes time as well as joint effort of several departments in the hospital to prepare the SEDs, causing considerable waiting time for the patient. Further, the use of allogeneic drops allows immediate access to SEDs in case time is limited to prevent corneal scars, ulcers, infiltrates or even transplants, epithelial defects or low vision due to epithelial surface disease.

Allogeneic SEDs are derived from healthy donors and are produced by a blood bank facility. Blood banks are experienced and equipped to produce blood products in a good manufacturing practice (GMP) environment. They can perform quality control, and are able to produce larger quantities that are quickly available. For our study, donors with blood group AB will be selected to ensure ABO compatibility. Donors are further selected to be males that never had a blood transfusion to minimize anti-HLA titers.

No prospective double blind randomized cross-over trials are known to exist to detect a difference in result between the effect of allogeneic SED or autologous SED for ocular surface disease. This pilot study is intended to obtain insight in the ability of autologous and allogeneic SEDs to improve patient dry eye sensation. Our hypothesis is that autologous SEDs (in a 1:1 dilution with saline) result in an improvement of the patient dry eye sensation, while allogeneic SEDs (in a 1:1 dilution with saline) do not.

ELIGIBILITY:
Inclusion Criteria:

* chronic dry eye syndrome
* age 18 or higher
* expected to benefit from SEDs
* can donate sufficient blood to prepare autologous SEDs
* meet the donor guidelines of Sanquin (except for age, donation frequency and hemoglobin concentration)

Exclusion Criteria:

* has corneal lesions more than punctates
* has a history of unstable Herpes simplex virus (HSV) keratitis or is treated for HSV keratitis
* currently already uses SEDs
* pregnancy, lactating, or intending the become pregnant in the next 3 months
* unable or unwilling to give informed consent
* active (systemic) microbial infection
* immuno-deficiency
* poor venous access

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2017-06-26 (Actual); Primary Completion 2018-10-08 (Actual); Study Completion 2018-10-08 (Actual)

PRIMARY OUTCOMES:
Ocular Surface Disease Index (OSDI) | One month after starting with serum eye drops
  Normalized OSDI score

SECONDARY OUTCOMES:
Tear production (Schirmer's test) | One month after starting with serum eye drops
  Millimeter
Tear break up time | One month after starting with serum eye drops
  Number of seconds before a dry spot appears in the tear film
Corneal punctates | One month after starting with serum eye drops
  Number

CONTACTS AND LOCATIONS:
Overall Officials: Pieter F van der Meer, PhD, Study Chair — Senior Scientist
Locations (1):
- Radboudumc, Nijmegen, Netherlands

IPD SHARING:
Plan to Share IPD: No